CLINICAL TRIAL: NCT03017339
Title: Effect of a Functional Exercise Program Associated With Low Level Laser Therapy on Pain, Functional Capacity and Quality of Life in Individuals With Fibromyalgia: A Double-blind Randomized Clinical Trial
Brief Title: Effect of a Functional Exercise Program Associated With Low Level Laser Therapy on Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Wouber Hérickson de Brito Vieira, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.442.759
Record Dates: First submitted 2017-01-04; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Fibromyalgia
Keywords: Low Lever Laser Therapy; Exercise Therapy; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser Group (Experimental): The subjects participated in a functional exercise program associated with low level laser therapy applied in the quadriceps, hamstrings and triceps sural
  Interventions: Other: Functional Exercise; Radiation: Low Level Laser Therapy
- Placebo Group (Placebo Comparator): The subjects participated in a functional exercise program associated with placebo low level laser therapy applied in the quadriceps, hamstrings and triceps sural
  Interventions: Other: Functional Exercise; Radiation: Placebo Low Level Laser Therapy

INTERVENTIONS:
Other: Functional Exercise
Radiation: Low Level Laser Therapy
  Arms: Laser Group
Radiation: Placebo Low Level Laser Therapy — Low Level Laser Therapy with the device off
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to investigate the effects of a functional exercise program associated with Low Level Laser Therapy (LLLT) on pain, functional capacity and quality of life of individuals with fibromyalgia. Half of participants will receive functional exercise and LLLT, while the other half will receive functional exercise and placebo LLLT.

ELIGIBILITY:
Inclusion Criteria:

* being female;
* age between 30 and 50 years;
* have an ovulatory cycle;
* height between 1.50m and 1.80m, body mass between 50 and 80 kg and BMI in the range of 18.5 to 29.9 kg / m2;
* present a clinical diagnosis of fibromyalgia, signed by a rheumatologist according to the current criteria of the American College of Rheumatology;
* is at least 6 months without any physical exercise;
* do not present musculoskeletal conditions that prevent them from performing the evaluation and proposed physical activity, except FM;
* not having diabetes mellitus and uncontrolled blood pressure;
* they do not present an inflammatory rheumatic condition or serious cardiovascular and / or pulmonary disease that prevents them from performing the evaluation and the proposed physical activity;
* Not having psychiatric illness or having malignant tumors;
* is not pregnant
* did not present dengue, zika or chikungunya in the last year;
* and finally not to be hypersensitive to light.

Exclusion Criteria:

* not attend for more than two consecutive exercise sessions
* at any time and for any reason expressing an intention to leave the study
* present a health problem that prevents them from continuing to carry out the proposed exercises

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain assessed by Visual Analogue Scale | Pain assessment two months after the intervention
  Assessed by Visual Analogue Scale
Pain assessed by Widespread Pain Index | Pain assessment two months after the intervention
  Assessed by Widespread Pain Index

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil